CLINICAL TRIAL: NCT05919797
Title: Association of Genetic Variations and Weight Loss Response to Naltrexone/Bupropion
Brief Title: Weight Loss Study: Genetics and Response to Naltrexone/Bupropion
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Judith Korner, Professor of Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAU3131; R01DK132527 (NIH)
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: Obesity; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Naltrexone-Bupropion combination; bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): Calorie restricted diet and treatment with Naltrexone/Bupropion
  Interventions: Drug: Naltrexone-Bupropion Combination

INTERVENTIONS:
Drug: Naltrexone-Bupropion Combination — Participants receive 28 weeks of naltrexone-bupropion weight loss medication during phase two of this study.
  Other Names: Contrave

SUMMARY:
The goal of this clinical trial is to understand if genetic variations are associated with the amount of weight loss with diet and while taking an FDA-approved medication for weight loss. The main question[s] it aims to answer are:

* In Aim One, the investigators propose to rigorously test the hypothesis that presence of the Taq1A A1+ polymorphism is associated with greater weight loss with NB compared with the A1- genotype.
* In Aim Two, the investigators will explore other genetic polymorphisms that might influence the efficacy of NB such as the fat mass and obesity-associated (FTO) gene which modulates DRD2 signaling, as carriers of risk alleles in both the FTO and ANKK1 gene demonstrate altered responses to reward-learning tasks associated with negative outcomes.

Participants will be in the study for 40 weeks, which consists of two phases:

1. From baseline to week 12, participants will receive individual nutritional counseling on a calorie restricted diet. This phase includes in-person visits, blood tests, an EKG, vital signs, questionnaires, body weight, and nutritional visits.
2. From week 12 to week 40, participants will continue to receive dietary counseling and will receive treatment with naltrexone/bupropion for 28 weeks. This phase includes in-person and phone visits, blood tests, vital signs, questionnaires, body weight, and nutritional visits.

DETAILED DESCRIPTION:
Weight loss can improve or prevent many obesity-related co-morbidities, yet time and again the cornerstone of obesity therapy - diet, physical activity and behavioral modification - fails to produce sufficient long-term weight loss in most individuals. In such cases, clinical guidelines recommend the addition of anti-obesity medication (AOM) when conservative methods are less than optimal. Yet even with the use of AOM, there is a wide range of inter-individual weight loss suggesting that there are "responders" and "non-responders." The variability in response to AOMs underscores the heterogeneity of obesity and the need for more personalized treatment that accounts for individual differences in etiologic factors. Given the strong heritability of obesity, it is possible that genetic factors play a role in an individual's response to a given pharmacotherapy.

This proposal focuses on the FDA-approved AOM, Contrave, which is a combination of two medications, naltrexone 32 mg and bupropion 360 mg (NB). Naltrexone is a µ-opioid receptor (MOPR) antagonist and bupropion inhibits the reuptake of dopamine and norepinephrine. Clinical trials of NB demonstrate a mean weight loss of 6.1% after 56 weeks of treatment; however, only 48% of patients achieved a clinically significant reduction in body weight of at least 5%. Knowledge of the likely mechanisms of action of NB makes it possible to address what might underlie the variability in response. The bupropion component of NB activates the proopiomelanocortin (POMC) neuron, a key regulator in decreasing food intake and stimulating energy expenditure, through stimulation of dopamine D2 receptors (DRD2). Naltrexone also activates POMC neurons by binding MOPR.

The investigators postulated that some of the variability in response to NB may be due to the Taq1A genetic variant (rs1800497) located in the ankyrin repeat and kinase domain-containing protein 1 (ANKK1) gene, adjacent to the DRD2 gene. Individuals carrying at least one minor allele of the rs1800497 polymorphism (termed Taq1A A1+) represent about 45% of the population and have 30-40% fewer brain DRD2. Carriers of the minor allele likely have a relative deficiency in dopaminergic activation of POMC neurons and, therefore, might receive the greatest benefit from a drug that activates POMC neurons. With this hypothesis in mind, the investigators conducted a retrospective proof-of-concept pilot study reviewing charts of patients treated with NB and found that individuals with the Taq1A A1+ genotype had a greater response compared with non-carriers, suggesting that this genotype could be used to predict successful weight loss.

In Aim One, the investigators propose to rigorously test the hypothesis that presence of the Taq1A A1+ polymorphism is associated with greater weight loss with NB compared with the A1- genotype. In Aim Two, the investigators will explore other genetic polymorphisms that might influence the efficacy of NB such as the fat mass and obesity-associated (FTO) gene which modulates DRD2 signaling, as carriers of risk alleles in both the FTO and ANKK1 gene demonstrate altered responses to reward-learning tasks associated with negative outcomes. Functional polymorphisms within genes that influence the metabolism of bupropion and naltrexone will also be examined in relation to weight loss outcomes. The ultimate goal is to incorporate pharmacogenetics into obesity medicine in order to maximize positive results and limit unnecessary cost and exposure to side effects of medications that provide minimal benefit to the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-65 years
* BMI 30-50 kg/m2 or
* BMI 27-29.99 kg/m2 with at least one weight-related comorbidity including controlled hypertension, dyslipidemia, obstructive sleep apnea, or osteoarthritis of a weight-bearing joint.

Exclusion Criteria:

* Obesity of known endocrine or hypothalamic origin
* HbA1c > 6.5%
* Cerebrovascular, cardiovascular, hepatic or renal disease
* History of seizures, serious psychiatric illness or suicide attempts, drug or alcohol misuse within prior 24 months
* Glaucoma
* Current tobacco use on a regular basis
* Use of dopamine agonists, opioid analgesics, antipsychotics, antidepressants, neuroleptics, naltrexone, diabetes medications
* Use of Monoamine oxidase (MAO) inhibitors < 14 days prior to screening
* Concomitant use of CYP2B6 inhibitors
* History of anorexia nervosa or bulimia
* Previous surgery for obesity
* Weight loss device intervention within prior 2 years
* Currently pregnant or lactating, planning pregnancy or refusal to use birth control when appropriate (Women of childbearing potential will be required to use effective contraception.)
* Blood pressure > 145/95 (use of anti-hypertensives will be allowed with the exception of verapamil, which can cause hyperprolactinemia)
* Clinically significant thyroid disease
* Triglycerides > 499 mg/dl
* Current use or use of weight loss medication within prior six months
* Any lifetime weight change deemed significant by Principal Investigator
* An affirmative answer to any question in the Columbia-Suicide Severity Rating Scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Percent Weight Loss (40 Weeks) | Baseline and 40 Weeks
  Percent weight loss from baseline to 40 weeks.

SECONDARY OUTCOMES:
Percent Excess Weight Loss | Baseline and 40 Weeks
  Percent excess weight loss defined as [(initial weight - weight lost at week 40)/(initial weight - weight at a BMI 25kg/m2)] x 100
Percent Excess Weight Loss | 12 Weeks and 40 Weeks
  Percent excess weight loss defined as [(Week 12 weight - weight lost at week 40)/(initial weight - weight at a BMI 25kg/m2)] x 100
Percent of Participants Achieving ≥ 5% Weight Loss | Baseline and 40 Weeks
  Percent of participants achieving ≥ 5% weight loss at week 40
Percent of Participants Achieving ≥ 10% Weight Loss | Baseline and 40 Weeks
  Percent of participants achieving ≥ 10% weight loss at week 40
Percent Weight Loss | 12 weeks and 40 weeks
  Percent weight loss from 12 weeks to 40 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Korner, MD,PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No